CLINICAL TRIAL: NCT00071409
Title: A Randomized, Double-blind, Placebo-controlled, Rising Dose, Multicenter Study to Evaluate the Efficacy and Safety of 90 Days of 300 or 600 mg Daily Subcutaneous Injections of INGAP Peptide in Type I Diabetes Mellitus Patients
Brief Title: Safety and Efficacy of INGAP-Peptide in Patients With Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Exsulin Corporation (Industry)
Responsible Party: Muhammad Rehman, MD, Procter and Gamble Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2003068
Record Dates: First submitted 2003-10-22; First posted 2003-10-23 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2011-08

CONDITIONS: Diabetes Mellitus, Insulin-Dependent
Keywords: Type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — INGAP peptide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- placebo (Placebo Comparator): 1.5 mL SC injection
  Interventions: Drug: placebo
- 300 mg INGAP Peptide (Experimental): 1.5 mL SC injection, once daily for 90 days
  Interventions: Drug: INGAP-Peptide
- 600 mg INGAP Peptide (Experimental): 1.5 mL SC injection, once daily for 90 days
  Interventions: Drug: INGAP-Peptide

INTERVENTIONS:
Drug: INGAP-Peptide — 1.5 mL, once daily, self-administered SC injection for 90 days
  Arms: 300 mg INGAP Peptide
Drug: INGAP-Peptide — 1.5 mL, once daily, self-administered SC injection for 90 days
  Arms: 600 mg INGAP Peptide
Drug: placebo — 1.5 mL, once daily, self-administered SC injection for 90 days
  Arms: placebo

SUMMARY:
Insulin is a chemical that the body needs in order to use or store sugar. It is made by a type of cell called a beta cell which resides in an organ known as the pancreas. Type 1 diabetes is a disease where the beta cells have been destroyed so that little or no insulin is made. Sugar levels rise in the blood as a result. INGAP-Peptide is being tested to attempt to create new beta cells in the pancreas, and to restore the ability to produce insulin in type 1 diabetic patients.

ELIGIBILITY:
Inclusion Criteria

* Age 18-65
* fasting C-peptide <0.3 ng/ml.
* HbA1c <10%
* history of onset of type 1 DM at or before 20 years of age.
* Otherwise healthy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2003-10; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
assess efficacy and safety based on arginine stimulated C peptide, fasting C peptide, average daily insulin dose, fasting glucose, glycosylated hemoglobin (Hb A1c), and AEs | 90 days

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Radiant Research, Irvine, California
  - VA Hospital UCSD, San Diego, California
  - Diablo Clinical Research, Walnut Creek, California
  - MedStar Clinical Research Center, Washington D.C., District of Columbia
  - Springfield Diabetes and Endocrine Center, Springfield, Illinois
  - Mercury Street Medical, Butte, Montana
  - UNC Diabetes Care Center, Durham, North Carolina
  - Clinical Research Institute of Southern Oregon, Medford, Oregon
  - University of Texas Health Science Center - Texas Diabetes Institute, San Antonio, Texas
  - DGD Research Associates, San Antonio, Texas